CLINICAL TRIAL: NCT01715402
Title: Optimization of Health Expenditure in Major Surgery: Impact of a Mixed, Clinical and Ethnographic Approach in the Model of Liver Surgery
Brief Title: Optimization of Health Expenditure in Liver Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 11060
Record Dates: First submitted 2012-10-22; First posted 2012-10-29 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Hepatocellular Carcinoma; Hilar Cholangiocarcinoma; Intra Hepatic Cholangiocarcinoma; Liver Metastasis
Keywords: liver tumor; carcinoma; cholangiocarcinoma; metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Klatskin Tumor; Carcinoma; Cholangiocarcinoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- operated patients: this cohort includes patients who underwent a liver surgery whatever the pathology and whatever the surgical procedure
  Interventions: Procedure: liver surgery

INTERVENTIONS:
Procedure: liver surgery — this intervention type includes hepatectomies; wedge; segmentectomies etc...

SUMMARY:
The aim of this study is to reduce the length of stay after liver surgery by taking account of objective quantitative clinical variables, subjective qualitative clinical variables and non clinical variables.

DETAILED DESCRIPTION:
a new dimension of the activity expected of physicians is to improve the safety of care on the one hand and the control of health care costs on the other.

key measures to help them are the publication of national recommendations, assessment of actual practices and the incentive to activity.

Internationalwide recent and concordant data suggest that

* quality and security of care, after an initial improvement, are going to stall
* scientific recommendations are rarely validated by an impact analysis and are not applied
* clinical data collected within an administrative framework are unreliable and too generalist
* the evaluation, especially in the surgical field, is based on indicators sometimes irrelevant and often unclear

ELIGIBILITY:
Inclusion Criteria:

* elective liver surgery
* older than 18
* agreed to participate
* surgical procedure included procedures registered as "HLFA003 - 007 ; 009 - 011 ; 017 - 020 ; HLFC002 à 004 ; 027 ; 032 ; 037" in the PMSI database

Exclusion Criteria:

* emergency surgery
* refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the population corresponds to patients operated in one of the thirteen hospitals.
  These hospitals are distributed on the french territory to ensure that the recruitment is representative of the general population
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
overall postoperative length of stay | during the 3 months after the surgery
  the overall postoperative length of stay is defined as the hospitalization between the surgery and patient's discharge.
  This period includes the readmission for at least 24 hours in case of outcomes related to the surgery.

SECONDARY OUTCOMES:
peroperative outcomes | during the surgical procedure
  the peroperative outcomes are collected during the surgery and correspond to any event occured during the surgical intervention
postoperative outcomes | after the surgery until postoperative month 3
  the postoperative outcomes correspond to any event occured after the surgical intervention. These outcomes include fistulae; bleeding...
construct of pronostic models | after the postoperative month 3
  the construct of pronostic models include variables that affect the length of stay; morbidity and mortality
evaluation of PMSI indicators | after the postoperative month 3
  this evaluation includes the analysis of PMSI indicators; their validity and the influence of centres on hepatectomies results

CONTACTS AND LOCATIONS:
Overall Officials: Olivier FARGES, MD, phD, Principal Investigator — Beaujon University Hospital
Locations (11):
- France (11):
  - Amiens North Hospital, Amiens
  - Bordeaux Hospital, Bordeaux
  - Beaujon University Hospital, Clichy
  - Lille Regional Hospital, Lille
  - Lyon Hospital, Lyon
  - Marseille Hospital, Marseille
  - Paoli calmette institute, Marseille
  - Saint Antoine Hospital, Paris
  - Strasbourg hospital, Strasbourg
  - Gustave Roussy institute, Villejuif
  - Paul Brousse Hospital, Villejuif

REFERENCES:
- [Derived] Cauchy F, Farges O, Vibert E, Boleslawski E, Pruvot FR, Regimbeau JM, Mabrut JY, Scatton O, Adham M, Laurent C, Gregoire E, Delpero JR, Bachellier P, Soubrane O. Sensitizing Surgeons to Their Outcome Has No Measurable Short-term Benefit. Ann Surg. 2017 Nov;266(5):884-889. doi: 10.1097/SLA.0000000000002403. PMID 28991876